CLINICAL TRIAL: NCT02783378
Title: 48 Hoursesophagal pH-monitoring With and Without Gaviscon
Brief Title: 48 Hours Esophagal pH-monitoring With and Without Gaviscon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Yvan Vandenplas, Prof. Dr, Universitair Ziekenhuis Brussel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: B.U.N. 143201627026
Record Dates: First submitted 2016-05-13; First posted 2016-05-26 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Gastroesophageal Reflux
Keywords: impedance metry; gaviscon
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gaviscon syrup (Other): Gaviscon will be given to threat patients with reflux after first 24 hours of oesophagal pH-monitoring.
  This is a syrup and will be given after every meal. dosage depends from age between 1ml and 5ml after every meal
  Interventions: Drug: Gaviscon Syrup

INTERVENTIONS:
Drug: Gaviscon Syrup
  Other Names: natriumalginaat and natriumbicarbonaat; BE386802.

SUMMARY:
At a esophagal pH-monitoring will the classic 24-hour measurement be extended to 48 hours. During the first 24 hours are the measurements without medication. After 24 hours the treatment will be started with Gaviscon and will the next 24 hours the measurements under the medication happen. Normally is the medication required after the measurements. With this study the investigators will have multiple measurement points to compare.

DETAILED DESCRIPTION:
This is an interventional, with questionnaires. 25 participants will be included.

Parents and children must be willing to have the esophagal pH-monitoring for 48 hours instead of 24 hours.

The restrictions are (like any other esophagal pH-monitoring) :

Do not detach the probe, no bath or shower, no bouncy castle, no swimming pool, ....

Give your child time to get used to the probe. Give your child no carbonated beverages, limit sweets, avoid chewing gum!

Not study specific procedures : there will be placed a probe for the oesophagal pH-monitoring and this will be checked on children's radiology.

study specific procedures : questionnaires at specific times : Before start : SF 36 Every 6 hours during 48hours : FLACC Satisfaction scale at the start, after 1 day and after 2 days

Flowchart time 0: obtaining ICF, signed by both parents, placing of probe, explanation of questionnaires, completing SF36 and satisfaction scale time 6: FLACC time 12: FLACC time 18: FLACC time 24: FLACC, satisfaction scale, reading out pH monitoring from the first 24 hours, then starting of Gaviscon in function of the result. The Gaviscon is supplied by the service, at no cost to the patient time 30: FLACC time 36: FLACC time 42: FLACC time 48: FLACC, satisfaction scale, remove pH monitoring

Calculation of the number of participants :

since there is never such a study was carried out, we started this pilot study. An analysis will be carried out after 15 patients.

Analysis of the results :

the results of the first and second 24 hour data will be compared (automatically by computer analysis).

ELIGIBILITY:
Inclusion Criteria:

* children in whom a pH-monitoring was asked
* pre school-age children
* hospitalized children
* parents have the informed consent signed.

Exclusion criteria :

* children over 6 years

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2016-02-24 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of pathological GERD | 24 and 48 hours
  change in pathological GERD from baseline at 24 and 48 hours

SECONDARY OUTCOMES:
Effect of Gaviscon on pain in infants with GERD | 24 and 48 hours
  Pain assessed via FLACC scale
Effect of Gaviscon on parental concern for parents of infants with GERD | 24 hours and 48 hours
  Parental concern assessed via 10 point Likert scale

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided